CLINICAL TRIAL: NCT02992184
Title: PoC-HCV Genedrive Viral Detection Assay Validation Study
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: EPISTEM (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANRS HC POC VIRAL DETECTION
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Hepatitis C
Keywords: HCV; Genedrive; Point of Care
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCV patients: 228 HCV patients
  Interventions: Device: HCV RNA detection with Genedrive assay; Device: HCV RNA detection with RealTime HCV
- control: 189 controls
  Interventions: Device: HCV RNA detection with Genedrive assay; Device: HCV RNA detection with RealTime HCV

INTERVENTIONS:
Device: HCV RNA detection with Genedrive assay
  Other Names: HCV RNA detection with Point of Care assay
Device: HCV RNA detection with RealTime HCV
  Other Names: HCV RNA detection with RT-PCR assay

SUMMARY:
The principal objective is to assess the diagnostic accuracy of the PoC assay (Genedrive, Epistem) to detect HCV RNA against the reference standard of commercial real-time polymerase chain reaction (RT-PCR) assay (RealTime HCV, Abbott) using stored heparinized plasma from patients with chronic hepatitis C and non-infected controls.

ELIGIBILITY:
Inclusion Criteria:

Criteria for case

* Age > 18 years old.
* Patients with positive HCV RNA.
* Heparinized plasma samples are available before the initiation of antiviral HCV therapy.
* Patients have given a written consent that their blood samples will be further used for research.

Criteria for control

* Age > 18 years old.
* Participants were tested negative for anti-HCV antibody
* Heparinized plasma samples are available
* Participants have given a written consent that their blood samples will be further used for research

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre-treatment cohort: 228 HCV patients samples
  * Age > 18 years old.
  * Patients with positive HCV RNA.
  * Heparinized plasma samples are available before the initiation of antiviral HCV therapy.
  * Patients have given a written consent that their blood samples will be further used for research.
  Control samples : 189 controls
  * Age > 18 years old.
  * Participants were tested negative for anti-HCV antibody
  * Heparinized plasma samples are available
  * Participants have given a written consent that their blood samples will be further used for research
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of HCV RNA detection with PoC assay (Genedrive, Epistem) vs reference standard of commercial real-time polymerase chain reaction (RT-PCR) assay (RealTime HCV, Abbott). | pre-treatment
  Assess the diagnostic accuracy of the PoC assay (Genedrive, Epistem) to detect HCV RNA against the reference standard of commercial real-time polymerase chain reaction (RT-PCR) assay (RealTime HCV, Abbott) using stored heparinized plasma from patients with chronic hepatitis C and non-infected controls (with Genedrive channel acceptance set at 2 out of 3).

SECONDARY OUTCOMES:
Diagnostic algorithm optimization | Pre-treatment
  To optimize the diagnostic algorithm (i.e., 1, 2, or 3 out of 3 channels; repeat testing or not) that gives the optimal balance between sensitivity and specificity for detection of HCV RNA.
Factors associated with false-positive of false-negative results | Pre-treatment
  To identify factors associated with false-positive or false-negative results of the PoC assay.
Assess the inter-examiner reproducibility of the PoC assay. | Pre-treatment

REFERENCES:
- [Derived] Llibre A, Shimakawa Y, Mottez E, Ainsworth S, Buivan TP, Firth R, Harrison E, Rosenberg AR, Meritet JF, Fontanet A, Castan P, Madejon A, Laverick M, Glass A, Viana R, Pol S, McClure CP, Irving WL, Miele G, Albert ML, Duffy D. Development and clinical validation of the Genedrive point-of-care test for qualitative detection of hepatitis C virus. Gut. 2018 Nov;67(11):2017-2024. doi: 10.1136/gutjnl-2017-315783. Epub 2018 Apr 3. PMID 29615488